CLINICAL TRIAL: NCT03149081
Title: A "Window Trial" on Boswellia, an Extract From Frankincense, for Breast Primary Tumors
Brief Title: A "Window Trial" on Boswellia for Breast Cancer Primary Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102688
Record Dates: First submitted 2017-05-04; First posted 2017-05-11 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Frankincense

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Boswellia (Experimental): Boswellia will be given at 800mg by mouth three times a day, immediately after each meal. Boswellia will be given from the time surgical resection is scheduled until the night before surgical resection.
  Interventions: Drug: Boswellia

INTERVENTIONS:
Drug: Boswellia — Boswellia is an extract from frankincense

SUMMARY:
The purpose of this study is to determine whether oral administration of Boswellia causes biological changes in primary tumors of breast cancer patients.

DETAILED DESCRIPTION:
To determine whether oral administration of Boswellia serrata causes biological changes related to angiogenesis (CD31), apoptosis (DNA fragmentation), and cell proliferation (Ki67) in primary tumors of breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ductal carcinoma in situ (DCIS) or invasive breast cancer (stages I, II, or III) with primary tumor(s) ≥ 1.0 cm on mammogram, ultrasound, MRI, or physical exam
* 18 years of age or older
* Subject must understand risks and benefits of the protocol and be able to give informed consent
* Females of child-bearing potential must agree to use an approved form of birth control and to have a negative pregnancy test result before and throughout the study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic and end organ function
* Ability and capacity to comply with the study and follow-up procedure
* Subjects must be scheduled for surgery at MUSC no less than 5 days from the planned start of day 1 and no more than 56 days from the planned start of day 1.
* At least 6 sections of unstained slides should be obtained. If sufficient slides or tissue is unavailable, the patient will be excluded from the trial.

Exclusion Criteria:

* Subjects undergoing neoadjuvant chemotherapy or neoadjuvant endocrine therapy
* Subjects with end-stage kidney disease and/or grade II liver dysfunction
* Subject has active or history of deep vein thrombosis (DVT)
* Subject has a history of coagulopathies or hematological disorders
* Subjects who are pregnant or are lactating.
* Subjects already taking drugs known to be 5-lipoxygenase inhibitors (Refer to section 5)
* Subjects taking drugs that interact with OATP1B3 (an anion transporter), MRP2 (a multidrug resistant protein), and/or P-Glycoprotein (P-Gp) (Refer to section 5.)
* Subjects taking anti-coagulants or platelet inhibitors (Refer to section 5)
* Subjects with bowel obstruction
* Subjects undergoing emergency surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Change in tumor proliferation rate | up to 56 days
  Change in tumor proliferation rate will be based on Ki67, CD31 and TUNEL assays in biopsies pre and post treatment with boswellia

SECONDARY OUTCOMES:
Number of adverse events reported | up to 84 days
  Safety data will be tabulated by type and grade of adverse event and will use CTCAE v. 4.0
Changes in tumors analyzed through immunohistochemistry | up to 56 days
  Additional changes in tumors as a result of boswellia intake will be analyzed through immunohistochemistry on paraffin-embedded tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Klauber-DeMore, MD, FACS, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No